CLINICAL TRIAL: NCT03606122
Title: Evaluation of the Suitability of a 5-ALA Patch (PD P 506 A, Alacare®) in the Photodynamic Therapy (PDT) of Actinic Keratosis on the Upper Extremities
Brief Title: 5-ALA Patch-PDT of Actinic Keratosis on the Upper Extremities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK 13
Record Dates: First submitted 2018-07-11; First posted 2018-07-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-12

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratosis on the upper extremities
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD P 506 A-PDT (Experimental): The study medication will be applied to each study lesion for 4 hours. After removal of the study medication the study lesions will be illuminated with red light of defined wavelength (PDT). Second PDT of the lesions will be performed 6-14 days after the first PDT.
  Interventions: Drug: PD P 506 A

INTERVENTIONS:
Drug: PD P 506 A — PD P 506 A is a dermal patch of 4 cm² in size loaded with 2 mg 5-ALA (as 5-ALA HCl) per cm²
  Other Names: Alacare®

SUMMARY:
This study evaluates the potential usefulness of photodynamic therapy with PD P 506 A in patients with actinic keratosis on the upper extremities for the first time.

DETAILED DESCRIPTION:
Patients will receive a second PD P 506 A-PDT on all AK lesions 1-2 weeks after the first PDT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been signed prior to or at Screening Visit
* Caucasian male and female patients
* Age ≥ 18 years
* Diagnosis of actinic keratosis (AK) with at least three locally separated lesions located on the upper extremities
* Selected AK study lesions have clearly defined margins and are mild to severe (grades I to III):
* Mild grade (I): Slight palpability, better felt than seen
* Moderate grade (II): Moderately thick AK, easily felt
* Severe grade (III): Very thick and/or obvious AK
* Skin sun sensitivity type I to IV according to Fitzpatrick

Exclusion Criteria:

* PDT Non-responder
* Pre-treatment of the AK lesions eligible for study procedures with pharmaceuticals approved for the treatment of AK during the 4 weeks preceding PDT (e.g. antineoplastic topical formulations as e.g. Metvix®, Ameluz®, Luxerm®, Solaraze®, Aldara®, Picato®, Actikerall®, 5-FU or vitamin A acid containing formulations)
* Pre-treatment of the AK lesions eligible for study procedures during the 2 weeks preceding PDT with keratolytic agents e.g. TCA, urea or salicylic acid containing formulations
* Pre-treatment with hypericin during the 2 weeks preceding PDT
* Treatment with systemic retinoids during the 3 months preceding PDT
* Treatment with cytostatics or radiation during the 3 months preceding PDT
* Female patients of childbearing potential (A female is considered of childbearing potential unless she has had tubal ligation, hysterectomy or has been postmenopausal, i.e. with spontaneous amenorrhea for at least 12 months.)
* Patients with clinically relevant suppression of the immune system
* Diagnosis of Porphyria
* Known photodermatoses of varying pathology and frequency, e.g. metabolic disorders such as aminoaciduria, idiopathic or immunological disorders such as polymorphic light reaction, genetic disorders such as xeroderma pigmentosum, and diseases precipitated or aggravated by exposure to sun light such as lupus erythematosus or pemphigus erythematosus
* Concomitant use of medicinal products with known phototoxic or photoallergic potential such as hypericin, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones and tetracyclines
* Skin diseases that might interfere with response evaluation of study PDT
* Skin sun sensitivity type V or VI according to Fitzpatrick
* Known intolerance to one or more of the ingredients of the study medication
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give a written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding inclusion
* Suspected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
The primary aim of the study is the evaluation of the clinical activity of PD P 506 A-PDT of AK on the upper extremities on lesion basis 12 weeks after treatment. | 12 weeks after treatment.
  Percentage of lesions with Clinically Complete Clearance (CCR) 12 weeks after two study treatments.

SECONDARY OUTCOMES:
Number and severity of treatment-related adverse events as assessed by NIA Adverse Event and Serious Adverse Event Guidelines. | 12 weeks after treatment.
  The secondary aim of the study is the evaluation of safety and tolerability of PD P 506 A-PDT of AK on the upper extremities.
In addition, the percentage of lesions with at least partial clearance 12 weeks after last study treatment will be analysed as a secondary parameter | 12 weeks after treatment.
  Percentage of lesions with at least partial clearance 12 weeks after two study treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Reinhold, Professor, Principal Investigator — Dermatologisches Zentrum Bonn
Locations (1):
- Dermatologisches Zentrum Bonn Friedensplatz, Bonn, Germany